CLINICAL TRIAL: NCT06370130
Title: Determation of Median Effective Dose of Propofol Combined With Different Dose of Esketamine Inhibiting Response to Laryngeal Mask Airway Insertion in Female Patients
Brief Title: Different Dose of Esketamine Inhibiting Response to Laryngeal Mask Airway Insertion
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Aerospace Center Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AerospaceCH
Record Dates: First submitted 2024-04-12; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Anesthesia
Keywords: Esketamine; propofol; median effective dose
MeSH Terms: interventions — Esketamine; Propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- K1 (Experimental): a group administered 0.2 mg/kg of esketamine
  Interventions: Drug: Esketamine 0.2mg/kg
- K2 (Active Comparator): a group administered esketamine of 0.3 mg/kg (K2)
  Interventions: Drug: Esketamine 0.3mg/kg

INTERVENTIONS:
Drug: Esketamine 0.2mg/kg — Patients received 0.2 mg/kg of esketamine intravenously for 30 s，after 120 s of propofol and disappearance of the eyelash reflex, a laryngeal mask was inserted.
  The test was performed using the sequential method. The initial dose of propofol was 2 mg/kg, which can be easily inserted into the LMA, and the propofol dose ratio of the adjacent patient was 0.9. If there was a positive reaction to the LMA insertion, the gradient was increased for the next patient; otherwise, the gradient was decreased, and the study was terminated after seven crossover inflection points.
  Other Names: propofol
  Arms: K1
Drug: Esketamine 0.3mg/kg — Patients received 0.3 mg/kg of esketamine intravenously for 30 s，after 120 s of propofol and disappearance of the eyelash reflex, a laryngeal mask was inserted.
  The test was performed using the sequential method. The initial dose of propofol was 2 mg/kg, which can be easily inserted into the LMA, and the propofol dose ratio of the adjacent patient was 0.9. If there was a positive reaction to the LMA insertion, the gradient was increased for the next patient; otherwise, the gradient was decreased, and the study was terminated after seven crossover inflection points.
  Other Names: propofol
  Arms: K2

SUMMARY:
Objective To prospectively determine the median effective dose (ED50) of propofol for inhibiting a response to laryngeal mask airway (LMA) insertion when combined with different doses of esketamine in female patients.

Methods Fifty-eight female patients (aged 20-60, ASAⅠ-Ⅱ) scheduled for elective hysteroscopy were enrolled and randomly divided into two groups, one administered 0.2 mg/kg of esketamine (K1 group, n = 28) and the other 0.3 mg/kg of esketamine (K2 group, n = 30). The two groups received the corresponding doses of esketamine intravenously, followed by an intravenous injection of propofol (injection time was 30 s). The initial dose of propofol was 2 mg/kg, and the dose ratio of propofol in the adjacent patients was 0.9. If there was a positive reaction to LMA insertion, the dose ratio in the next patient was increased by one gradient, and if not, the dose ratio was decreased by one gradient. The median effective dose (ED50), 95% effective dose (ED95) and 95% confidence interval (95%CI) of propofol for inhibiting a response to LMA insertion in the two esketamine groups were calculated using a probit analysis.

ELIGIBILITY:
Inclusion Criteria:

* women undergoing gynaecological hysteroscopy and surgery resulting from any indication
* age: from 20 to 60 years old
* body mass index (BMI): 18-30 kg/m2
* American Society of Anesthesiologists Physical Status score: grade I-II
* voluntary participation in this study

Exclusion Criteria:

* pregnant and lactating women
* patients with a history of propofol allergy, uncontrolled hypertension, hyperthyroidism, severe cardiopulmonary diseases, airway stenosis and mental diseases
* those who have recently taken or are taking psychotropic drugs or analgesic drugs
* patients allergic to or addicted to esketamine

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2023-03-10 (Actual)

PRIMARY OUTCOMES:
Record of the patient response during LMA placement | 1 minutes
  body movement or no body movement. Body movement is defined as cough, breath-holding or laryngospasm when the LMA is inserted or the laryngeal cuff inflated, and the patient has difficulty opening the mouth and conscious movement all over the body. No body movement is defined as the absence of these reactions when the LMA is inserted or the laryngeal cuff is inflated.
Overall condition of LMA placement | 1 minutes
  mouth opening ≥3 cm is complete and <3 cm is incomplete. The LMA placement conditions are as follows: 1 = complete relaxation, 2 = mild resistance, 3 = resistance but can open the mouth, 4 = resistance and the need to further increase the propofol dose; 1 and 2 are considered successful LMA placement and 3 and 4 are failure
Record related indicators | 1 minutes
  Record of the mean arterial pressure (MAP)
Record related indicators | 2 minutes
  Record of the mean arterial pressure (MAP)
Record related indicators | 1 minutes
  heart rate (HR)
Record related indicators | 2minutes
  heart rate (HR)
Record of additional doses of propofol and the adverse reactions of positive patients during the induction process (hypotension, bradycardia and apnoea, etc.) | 1 minutes
  If the patient develops bradycardia (<45 beats/min), 0.3-0.5 mg of intravenous atropine is given, and 1-2 mg of intravenous dopamine is administered for hypotension (<20% of basal blood pressure)

CONTACTS AND LOCATIONS:
Locations (1):
- Liang-Yuan Lu, Beijing, Beijing Municipality, China